CLINICAL TRIAL: NCT04293562
Title: A Phase 3 Randomized Trial for Patients With De Novo AML Comparing Standard Therapy Including Gemtuzumab Ozogamicin (GO) to CPX-351 With GO, and the Addition of the FLT3 Inhibitor Gilteritinib for Patients With FLT3 Mutations
Brief Title: A Study to Compare Standard Chemotherapy to Therapy With CPX-351 and/or Gilteritinib for Patients With Newly Diagnosed AML With or Without FLT3 Mutations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAML1831; NCI-2020-00546 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML1831 (Other: Children's Oncology Group); AAML1831 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-02-18; First posted 2020-03-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Stem Cell Transplantation; asparaginase erwinia chrysanthemi recombinant; Asparaginase; Specimen Handling; Biopsy; Cytarabine; Daunorubicin; Dexrazoxane; Razoxane; Etoposide; Fluorodeoxyglucose F18; Gemtuzumab; gilteritinib; CPX-351; Injections; Liposomes; Magnetic Resonance Spectroscopy; Methotrexate; merphos; Mitoxantrone; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Arm A High Risk Group (Experimental): Arm A High Risk Group: See Detailed Description.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm A Low Risk Group 1 (Experimental): Arm A Low Risk Group 1: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm A Low Risk Group 2 (Experimental): Arm A Low Risk Group 2: See Detailed Description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm AC High Risk Group (Experimental): Arm AC High Risk Group: See Detailed Description.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm AC Low Risk Group 2 (Experimental): Arm AC Low Risk Group 2: See Detailed Description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm AD High Risk Group (Experimental): Arm AD High Risk Group: See Detailed Description.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm AD Low Risk Group 2 (Experimental): Arm AD Low Risk Group 2: See Detailed Description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm B High Risk Group (Experimental): Arm B High Risk Group: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm B Low Risk Group 1 (Experimental): Arm B Low Risk Group 1: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm B Low Risk Group 2 (Experimental): Arm B Low Risk Group 2: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm BC High Risk Group (Experimental): Arm BC High Risk Group: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm BC Low Risk Group 2 (Experimental): Arm BC Low Risk Group 2: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm BD High Risk Group (Experimental): Arm BD High Risk Group: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone
- Arm BD Low Risk Group 2 (Experimental): Arm BD Low Risk Group 2: See Detailed Description. (CLOSED TO ACCRUAL 11/19/2024)
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Dexrazoxane Hydrochloride; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Gemtuzumab Ozogamicin; Drug: Gilteritinib Fumarate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
  Arms: Arm A High Risk Group; Arm AC High Risk Group; Arm AD High Risk Group; Arm B High Risk Group; Arm BC High Risk Group; Arm BD High Risk Group
Drug: Asparaginase Erwinia chrysanthemi — Given IM or IV
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
  Arms: Arm A Low Risk Group 1; Arm A Low Risk Group 2; Arm AC Low Risk Group 2; Arm AD Low Risk Group 2; Arm B Low Risk Group 1; Arm B Low Risk Group 2; Arm BC Low Risk Group 2; Arm BD Low Risk Group 2
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo BM aspiration
Procedure: Bone Marrow Biopsy — BM biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cytarabine — Given IV or IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Arm A High Risk Group; Arm A Low Risk Group 1; Arm A Low Risk Group 2; Arm AC High Risk Group; Arm AC Low Risk Group 2; Arm AD High Risk Group; Arm AD Low Risk Group 2
Drug: Dexrazoxane Hydrochloride — Given IV
  Other Names: Cardioxane; Totect; Zinecard
  Arms: Arm A High Risk Group; Arm A Low Risk Group 1; Arm A Low Risk Group 2; Arm AC High Risk Group; Arm AC Low Risk Group 2; Arm AD High Risk Group; Arm AD Low Risk Group 2; Arm BC Low Risk Group 2; Arm BD Low Risk Group 2
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Other: Fludeoxyglucose F-18 — Undergo FDG-PET
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Gilteritinib Fumarate — Given PO/NG/G-tube
  Other Names: ASP-2215 Hemifumarate; ASP2215 Hemifumarate; Gilteritinib Hemifumarate; Xospata
  Arms: Arm AC High Risk Group; Arm AC Low Risk Group 2; Arm AD High Risk Group; Arm AD Low Risk Group 2; Arm BC High Risk Group; Arm BC Low Risk Group 2; Arm BD High Risk Group; Arm BD Low Risk Group 2
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX 351; CPX-351; CPX351; Cytarabine and Daunorubicin Liposomal; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
  Arms: Arm B High Risk Group; Arm B Low Risk Group 1; Arm B Low Risk Group 2; Arm BC High Risk Group; Arm BC Low Risk Group 2; Arm BD High Risk Group; Arm BD Low Risk Group 2
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Arm A High Risk Group; Arm A Low Risk Group 1; Arm A Low Risk Group 2; Arm AC High Risk Group; Arm AC Low Risk Group 2; Arm AD High Risk Group; Arm AD Low Risk Group 2; Arm B High Risk Group; Arm B Low Risk Group 1; Arm BC High Risk Group; Arm BC Low Risk Group 2; Arm BD High Risk Group; Arm BD Low Risk Group 2
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
  Arms: Arm A Low Risk Group 2; Arm AC Low Risk Group 2; Arm AD Low Risk Group 2; Arm B Low Risk Group 2; Arm BC Low Risk Group 2; Arm BD Low Risk Group 2
Procedure: Positron Emission Tomography — Undergo FDG-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid

SUMMARY:
This phase III trial compares standard chemotherapy to therapy with liposome-encapsulated daunorubicin-cytarabine (CPX-351) and/or gilteritinib for patients with newly diagnosed acute myeloid leukemia with or without FLT3 mutations. Drugs used in chemotherapy, such as daunorubicin, cytarabine, and gemtuzumab ozogamicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. CPX-351 is made up of daunorubicin and cytarabine and is made in a way that makes the drugs stay in the bone marrow longer and could be less likely to cause heart problems than traditional anthracycline drugs, a common class of chemotherapy drug. Some acute myeloid leukemia patients have an abnormality in the structure of a gene called FLT3. Genes are pieces of DNA (molecules that carry instructions for development, functioning, growth and reproduction) inside each cell that tell the cell what to do and when to grow and divide. FLT3 plays an important role in the normal making of blood cells. This gene can have permanent changes that cause it to function abnormally by making cancer cells grow. Gilteritinib may block the abnormal function of the FLT3 gene that makes cancer cells grow. The overall goals of this study are, 1) to compare the effects, good and/or bad, of CPX-351 with daunorubicin and cytarabine on people with newly diagnosed AML to find out which is better, 2) to study the effects, good and/or bad, of adding gilteritinib to AML therapy for patients with high amounts of FLT3/ITD or other FLT3 mutations and 3) to study changes in heart function during and after treatment for AML. Giving CPX-351 and/or gilteritinib with standard chemotherapy may work better in treating patients with acute myeloid leukemia compared to standard chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare event-free survival (EFS) in children with de novo acute myeloid leukemia (AML) without FLT3 mutations who are randomly assigned to standard induction therapy on Arm A with daunorubicin, cytarabine (DA) and gemtuzumab ozogamicin (GO) (DA-GO) versus Arm B with CPX-351 and GO.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) and rates of end of Induction 1 (EOI1) minimal residual disease (MRD) in children with de novo AML without FLT3 mutations who are randomly assigned to standard induction therapy (Arm A) with DA-GO versus CPX-351 and GO (Arm B).

II. To estimate the EFS and rate of EOI1 MRD in FLT3 internal tandem duplication mutation positive patients (FLT3/ITD+; as defined by allelic ratio > 0.1) without favorable cytomolecular characteristics (NPM1 and/or CEBPA) receiving gilteritinib fumarate (gilteritinib) in combination with DA-GO (Arm AC).

III. To estimate the EFS and rate of EOI1 MRD in patients with non-ITD FLT3 activating mutations who receive backbone therapy (DA-GO or CPX-351 and GO) with gilteritinib (Arms AD and BD).

IV. To determine the feasibility of combining gilteritinib and DA-GO or CPX-351 and GO in patients with FLT3/ITD and FLT3/TKD mutations (Arm AC/Arm BC/Arm AD/Arm BD).

V. To compare EOI1 MRD and EFS in patients with FLT3/ITD AML+ (allelic ratio [AR] > 0.1) without favorable cytogenetic/molecular characteristics treated with DA-GO-gilteritinib versus (vs) CPX-GO-gilteritinib (Arm AC vs Arm BC).

VI. To compare the incidence of significant left ventricular systolic dysfunction (LVSD) in children with de novo AML without FLT3 mutations who are randomly assigned to standard induction therapy (Arm A) with DA-GO versus CPX-351 and GO (Arm B).

VII. To compare the changes in echocardiography-derived measures of cardiac function, including left ventricular ejection fraction (EF) and global longitudinal strain (GLS), throughout AML therapy in patients with low and high risk AML without FLT3 mutations receiving Arm A vs Arm B.

VIII. Determine if early changes in sensitive echocardiographic measures of cardiac function (i.e., post-Induction 1 decline in GLS) and elevations in circulating cardiac biomarkers (i.e., cardiac troponin T and N-terminal pro b-type natriuretic peptide) are associated with subsequent declines in left ventricular ejection fraction in patients with non-FLT3 mutant AML receiving therapy on Arms A or B.

IX. To compare longitudinal acute changes in neuropsychological functioning and neurocognitive late effects between those with central nervous system (CNS) disease and those without CNS disease and between those treated with hematopoietic stem cell transplant (HSCT) and those treated with chemotherapy only for patients on Arms A and B.

X. To compare cardiotoxicity measures (EF, GLS, and cardiac biomarkers) in patients receiving standard induction with dexrazoxane hydrochloride (dexrazoxane) vs. CPX-351 in the context of gilteritinib therapy and explore whether the differential cardiotoxicity across arms varies from that observed in non-FLT3 mutant AML without gilteritinib exposure.

EXPLORATORY OBJECTIVES:

I. To estimate the EFS and rate of EOI1 MRD in patients with high allelic ratio (HAR) FLT3/ITD+ patients, as historically defined by an AR > 0.4, receiving gilteritinib in combination with DA-GO (Arm AC with AR > 0.4).

II. To estimate the EFS, OS, and rate of EOI1 MRD in FLT3/ITD+ patients (as defined by allelic ratio > 0.1) with NPM1 and/or bZIP CEBPA mutations receiving gilteritinib in combination with DA-GO (Arm AC).

III. Compare the changes in high sensitivity troponin and natriuretic peptide elevations throughout AML therapy, as measured at the end of each chemotherapy course, in patients with low and high risk AML without FLT3 mutations receiving Arm A vs Arm B.

IV. Quantify the association of host factors (age, sex, body mass index [BMI], race), treatment exposures (cumulative anthracycline dose, anthracycline arm, hematopoietic stem cell transplant vs. chemotherapy alone), early declines in GLS, and elevations in cardiac biomarkers (cTnT and NT-proBNP) with subsequent LVSD.

V. To describe the rates of CNS disease utilizing an updated strategy for diagnosing and defining CNS disease in pediatric AML.

VI. To describe the rates of CNS relapse (both isolated CNS and combined bone marrow/CNS) when utilizing this updated strategy as well as changing CNS prophylaxis and treatment to include triple intrathecal chemotherapy.

VII. To describe the rate of bone marrow measurable residual disease, detected by multi-dimensional flow cytometry, prior to hematopoietic stem cell transplant (HSCT).

VIII. To describe plasma metabolomics that may impact efficacy, toxicity, and/or pharmacokinetics of allogeneic HSCT.

IX. To estimate the prevalence of non-risk stratifying cytogenetic/molecular variants and assess their impact on outcome in childhood AML.

X. To describe the pharmacokinetic parameters of plasma cytarabine and daunorubicin after CPX-351 administration to pediatric and young adult patients with new diagnosis of AML.

XI. To describe the pharmacokinetic parameters of orally administered gilteritinib when administered to pediatric and young adult patients with new diagnosis of AML.

XII. To describe the pharmacodynamic parameters of gilteritinib using the FLT3 plasma inhibitory activity assay (PIA) when administered to children and young adults with new diagnosis of AML and FLT3 mutations.

XIII. To estimate OS in patients with FLT3/ITD+ AML (AR > 0.1) without favorable cytogenetic/molecular characteristics treated with DA-GO-gilteritinib or CPX-351-GO-gilteritinib (Separate analyses will be conducted for Arm AC vs Arm BC).

OUTLINE: Patients are randomized to either Arm A or B and assigned to Arm C or D based on FLT3 testing results. As of 11/19/24 arms B, BC and BD are closed and new patients receive treatment in Arm A Low Risk Group 2 Induction 1 or Arm A High Risk Induction 1, and then assigned to arm AC or AD per FLT3 results.

Risk group assignments are calculated based on cytogenetic, molecular and genomic findings (details in protocol)

1. Low Risk 1
2. Low Risk 2
3. High Risk

   TREATMENT FOR PATIENTS WITHOUT FLT3 MUTATIONS:

   ARM A LOW RISK GROUP 1:

   INDUCTION 1: Patients receive cytarabine intravenously (IV) over 1-30 minutes every 12 hours (Q12H) on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS1 receive methotrexate intrathecally (IT), therapeutic hydrocortisone (hydrocortisone) IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT once weekly (QW) starting on day 8 for 4-6 weeks (may continue into Induction 2) until the cerebral spinal fluid (CSF) is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2: Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8 and dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5.

   INTENSIFICATION 1: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5.

   INTENSIFICATION 2: Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9. Patients also receive asparaginase Erwinia chrysanthemi intramuscularly (IM) on days 2 and 9 or IV over 1-2 hours on days 2 and 9.

   ARM B LOW RISK GROUP 1:

   INDUCTION 1: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2: Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5.

   INTENSIFICATION 1: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5.

   INTENSIFICATION 2: Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9. Patients also receive asparaginase Erwinia chrysanthemi IM on days 2 and 9 or IV over 1-2 hours on days 2 and 9.

   ARM A LOW RISK GROUP 2:

   INDUCTION 1: Patients receive cytarabine IV over 1-30 minutes Q12H on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2: Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8 and dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5.

   INTENSIFICATION 1: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5.

   INTENSIFICATION 2: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H on days 1-4 and dexrazoxane IV over 15 minutes and mitoxantrone hydrochloride (mitoxantrone) IV over 5-15 minutes on days 3-6.

   INTENSIFICATION 3: Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9. Patients also receive asparaginase Erwinia chrysanthemi IM on days 2 and 9 or IV over 1-2 hours on days 2 and 9.

   ARM B LOW RISK GROUP 2:

   INDUCTION 1: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2: Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5.

   INTENSIFICATION 1: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5.

   INTENSIFICATION 2: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H on days 1-4 and dexrazoxane IV over 15 minutes and mitoxantrone hydrochloride (mitoxantrone) IV over 5-15 minutes on days 3-6.

   INTENSIFICATION 3: Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9. Patients also receive asparaginase Erwinia chrysanthemi IM on days 2 and 9 or IV over 1-2 hours on days 2 and 9.

   ARM A HIGH RISK GROUP:

   INDUCTION 1: Patients receive cytarabine IV over 1-30 minutes Q12H on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2: Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8 and dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5.

   INTENSIFICATION 1: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5.

   HSCT: After completion of Intensification 1 and investigator assigned conditioning regimen, patients undergo allogeneic HSCT.

   ARM B HIGH RISK GROUP:

   INDUCTION 1: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 6. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2: Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5.

   INTENSIFICATION 1: Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5.

   HSCT: After completion of Intensification 1 and investigator assigned conditioning regimen, patients undergo allogeneic HSCT.

   TREATMENT FOR PATIENTS WITH FLT3/ITD MUTATIONS (ITD AR > 0.1):

   ARM AC LOW RISK GROUP 2:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive cytarabine IV over 1-30 minutes Q12H on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib orally (PO)/nasogastric (NG)/gastrostomy (G)-tube once daily (QD) on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO/NG/G-tube QD on days 6-26.

   INTENSIFICATION 2 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H on days 1-4, dexrazoxane IV over 15 minutes and mitoxantrone IV over 5-15 minutes on days 3-6, and gilteritinib PO/NG/G-tube QD on days 7-27.

   INTENSIFICATION 3 (WITH GILTERITINIB): Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9, asparaginase Erwinia chrysanthemi IM or IV over 1-2 hours, and gilteritinib PO/NG/G-tube QD on days 10-30.

   POST-CHEMOTHERAPY GILTERITINIB MAINTENANCE: Patients receive gilteritinib PO/NG/G-tube QD on days 1-365.

   ARM BC LOW RISK GROUP 2:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO/NG/G-tube QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5 and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO/NG/G-tube QD on days 6-26.

   INTENSIFICATION 2 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H on days 1-4, dexrazoxane IV over 15 minutes and mitoxantrone IV over 5-15 minutes on days 3-6, and gilteritinib PO/NG/G-tube QD on days 7-27.

   INTENSIFICATION 3 (WITH GILTERITINIB): Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9, asparaginase Erwinia chrysanthemi IM or IV over 1-2 hours, and gilteritinib PO/NG/G-tube QD on days 10-30.

   POST-CHEMOTHERAPY GILTERITINIB MAINTENANCE: Patients receive gilteritinib PO/NG/G-tube QD on days 1-365.

   ARM AC HIGH RISK GROUP:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive cytarabine IV over 1-30 minutes Q12H on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO/NG/G-tube QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO/NG/G-tube QD on days 6-26.

   HSCT: After completion of Intensification 1 and investigator assigned conditioning regimen, patients undergo allogeneic HSCT.

   POST-HSCT GILTERITINIB MAINTENANCE: Beginning 30-120 days after completion of HSCT, patients receive gilteritinib PO/NG/G-tube QD on days 1-365.

   ARM BC HIGH RISK GROUP:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO/NG/G-tube QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5 and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO/NG/G-tube QD on days 6-26.

   HSCT: After completion of Intensification 1 and investigator assigned conditioning regimen, patients undergo allogeneic HSCT.

   POST-HSCT GILTERITINIB MAINTENANCE: Beginning 30-120 days after completion of HSCT, patients receive gilteritinib PO/NG/G-tube QD on days 1-365.

   TREATMENT FOR NON-ITD FLT3 ACTIVATING MUTATIONS:

   ARM AD LOW RISK GROUP 2:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive cytarabine IV over 1-30 minutes Q12H on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO/NG/G-tube QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO/NG/G-tube QD on days 6-26.

   INTENSIFICATION 2 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H on days 1-4, dexrazoxane IV over 15 minutes and mitoxantrone IV over 5-15 minutes on days 3-6, and gilteritinib PO/NG/G-tube QD on days 7-27.

   INTENSIFICATION 3 (WITH GILTERITINIB): Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9, asparaginase Erwinia chrysanthemi IM or IV over 1-2 hours, and gilteritinib PO/NG/G-tube QD on days 10-30.

   POST-CHEMOTHERAPY GILTERITINIB MAINTENANCE: Patients receive gilteritinib PO/NG/G-tube QD on days 1-365.

   ARM BD LOW RISK GROUP 2:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO/NG/G-tube QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5 and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO/NG/G-tube QD on days 6-26.

   INTENSIFICATION 2 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H on days 1-4, dexrazoxane IV over 15 minutes and mitoxantrone IV over 5-15 minutes on days 3-6, and gilteritinib PO/NG/G-tube QD on days 7-27.

   INTENSIFICATION 3 (WITH GILTERITINIB): Patients receive high-dose cytarabine IV over 3 hours Q12H on days 1, 2, 8, and 9, asparaginase Erwinia chrysanthemi IM or IV over 1-2 hours, and gilteritinib PO/NG/G-tube QD on days 10-30.

   POST-CHEMOTHERAPY GILTERITINIB MAINTENANCE: Patients receive gilteritinib PO/NG/G-tube QD on days 1-365.

   ARM AD HIGH RISK GROUP:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive cytarabine IV over 1-30 minutes Q12H on days 1-10, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO/NG/G-tube QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive cytarabine IV over 1-30 minutes Q12H on days 1-8, dexrazoxane IV over 15 minutes and daunorubicin IV over 1-15 minutes on days 1, 3, and 5, and gilteritinib PO/NG/G-tube QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO QD on days 6-26.

   HSCT: After completion of Intensification 1 and investigator assigned conditioning regimen, patients undergo allogeneic HSCT.

   POST-HSCT GILTERITINIB MAINTENANCE: Beginning 30-120 days after completion of HSCT, patients receive gilteritinib PO or NG or G tube QD on days 1-365.

   ARM BD HIGH RISK GROUP:

   CONTINUED INDUCTION 1 (WITH GILTERITINIB): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, gemtuzumab ozogamicin IV over 2 hours on day 6, and gilteritinib PO QD on days 11-31. Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 8. Patients with CNS2, CNS3a, and CNS3b receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 8 for 4-6 weeks (may continue into Induction 2) until the CSF is clear of blasts (CNS1 status). Patients with CNS3c receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 1 for 6 weeks (may continue into Induction 2).

   INDUCTION 2 (WITH GILTERITINIB): Patients with CNS1 receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients with CNS2 receive methotrexate IT, hydrocortisone IT, and cytarabine IT QW starting on day 0 until CNS1 status is reached. Patients also receive CPX-351 IV over 90 minutes on days 1, 3, and 5 and gilteritinib PO QD on days 11-31.

   INTENSIFICATION 1 (WITH GILTERITINIB): Patients receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 0. Patients also receive high-dose cytarabine IV over 1-3 hours Q12H and etoposide IV over 90-120 minutes on days 1-5, and gilteritinib PO QD on days 6-26.

   HSCT: After completion of Intensification 1 and investigator assigned conditioning regimen, patients undergo allogeneic HSCT.

   POST-HSCT GILTERITINIB MAINTENANCE: Beginning 30-120 days after completion of HSCT, patients receive gilteritinib PO or NG or G tube QD on days 1-365.

   NOTE: During Induction 2 or Intensification 2, patients in Arms A and B with left ventricular systolic dysfunction receive a replacement course of high-dose cytarabine IV over 3 hours on days 1, 2, 8, and 9, and asparaginase Erwinia chrysanthemi IM or IV over 1-2 hours. Patients in Arms AC, BC, AD, and BD receive treatment as in Arms A and B and also receive gilteritinib PO QD on days 10-30 (Induction 2) or days 10-30 (Intensification 2).

   OPTIONAL NEUROCOGNITIVE STUDY:

   Patients may complete the Cogstate assessment battery at the end of Induction 1, at the end of therapy, and at 9 and 60 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be enrolled on APEC14B1 and consented to Eligibility Screening (Part A) prior to enrollment and treatment on AAML1831
* Patients must be less than 22 years of age at the time of study enrollment
* Patient must be newly diagnosed with de novo AML according to the 2016 World Health Organization (WHO) classification with or without extramedullary disease

  * Patient must have 1 of the following:

    * >= 20% bone marrow blasts (obtained within 14 days prior to enrollment)

      * In cases where extensive fibrosis may result in a dry tap, blast count can be obtained from touch imprints or estimated from an adequate bone marrow core biopsy
    * < 20% bone marrow blasts with one or more of the genetic abnormalities associated with childhood/young adult AML as provided in the protocol (sample obtained within 14 days prior to enrollment)
    * A complete blood count (CBC) documenting the presence of at least 1,000/uL (i.e., a white blood cell [WBC] count >= 10,000/uL with >= 10% blasts or a WBC count of >= 5,000/uL with >= 20% blasts) circulating leukemic cells (blasts) if a bone marrow aspirate or biopsy cannot be performed (performed within 7 days prior to enrollment)
* ARM C: Patient must be >= 2 years of age at the time of Late Callback
* ARM C: Patient must have FLT3/ITD allelic ratio > 0.1 as reported by Molecular Oncology
* ARM C: Patient does not have any congenital long QT syndrome or congenital heart block
* ARM C: Females of reproductive potential must agree to use effective contraception during treatment and for at least 6 months after the last dose of gilteritinib
* ARM C: Lactating women must agree not to breastfeed during treatment with gilteritinib and for 2 months after the last dose of gilteritinib
* ARM C: Males of reproductive potential must agree to use effective contraception during treatment and for at least 4 months after the last dose of gilteritinib
* ARM D: Patient must be >= 2 years of age at the time of Late Callback
* ARM D: Patient must have one of the clinically relevant non-ITD FLT3 activating mutations as reported by Foundation Medicine
* ARM D: Females of reproductive potential must agree to use effective contraception during treatment and for at least 6 months after the last dose of gilteritinib
* ARM D: Lactating women must agree not to breastfeed during treatment with gilteritinib and for 2 months after the last dose of gilteritinib
* ARM D: Males of reproductive potential must agree to use effective contraception during treatment and for at least 4 months after the last dose of gilteritinib
* NEUROPSYCHOLOGICAL TESTING: Patient must be enrolled on Arm A or Arm B. Patients who transfer to Arm C or Arm D are not eligible
* NEUROPSYCHOLOGICAL TESTING: Patient must be 5 years or older at the time of enrollment
* NEUROPSYCHOLOGICAL TESTING: English-, French- or Spanish-speaking
* NEUROPSYCHOLOGICAL TESTING: No known history of neurodevelopmental disorder prior to diagnosis of AML (e.g., Down syndrome, fragile X, William syndrome, mental retardation)
* NEUROPSYCHOLOGICAL TESTING: No significant visual or motor impairment that would prevent computer use or recognition of visual test stimuli
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Fanconi anemia
* Shwachman Diamond syndrome
* Patients with constitutional trisomy 21 or with constitutional mosaicism of trisomy 21
* Telomere disorders
* Germline predispositions known, or suspected by the treating physician to increase risk of toxicity with AML therapy
* Any concurrent malignancy
* Juvenile myelomonocytic leukemia (JMML)
* Philadelphia chromosome positive AML
* Mixed phenotype acute leukemia
* Acute promyelocytic leukemia
* Acute myeloid leukemia arising from myelodysplasia
* Therapy-related myeloid neoplasms
* Patients with persistent cardiac dysfunction prior to enrollment, defined as ejection fraction (EF) < 50% (preferred method Biplane Simpson's EF) or if EF unavailable, shortening fraction (SF) < 24%. *Note: if clinically safe and feasible, repeat echocardiogram is strongly advised in order to confirm cardiac dysfunction following clinical stabilization, particularly if occurring in the setting of sepsis or other transient physiologic stressor. If the repeat echocardiogram demonstrates an EF >= 50%, the patient is eligible to enroll and may receive an anthracycline-containing Induction regimen
* Administration of prior anti-cancer therapy except as outlined below:

  * Hydroxyurea
  * All-trans retinoic acid (ATRA)
  * Corticosteroids (any route)
  * Intrathecal therapy given at diagnosis
  * In particular, strong inducers of CYP3A4 and/or P-glycoprotein (P-gp) should be avoided from the time of enrollment until it is determined whether the patient will receive gilteritinib. Patients receiving gilteritinib will be required to avoid strong CYP3A4 inducers and/or strong P-gp inducers for the duration of the study treatment
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* ARM D: Patient does not have any congenital long QT syndrome or congenital heart block

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1186 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 3 years
  The Kaplan-Meier method will be used to estimate 3-year EFS, defined as the time from study entry until induction failure, relapse, secondary malignancy, or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years
  The Kaplan-Meier method will be used to estimate 3-year OS, defined as the time from study entry until death.
Proportion of patients positive for minimal residual disease (MRD+) | Up to 4 weeks
  The proportion of patients MRD+ at end of induction 1 (EOI1) will be estimated as the number of patients MRD+ divided by the number of patients with evaluable EOI1 MRD results along with a corresponding 95% confidence interval determined using a binomial exact method.
Proportion of patients who died during protocol therapy | Up to 2 years
  The proportion of patients who died during protocol therapy will be estimated along with the corresponding 95% confidence interval determined using a binomial exact method.
Incidence of adverse events | Up to 2 years
  The proportion of patients experiencing at least one grade 3 or higher non-hematologic toxicity and infection while on protocol therapy will be estimated along with the corresponding 95% confidence interval determined using a binomial exact method. Toxicity will be assessed by Common Terminology Criteria for Adverse Events version 5.0.
Relapse rate | Up to 3 years
  Cumulative incidence estimates will be used to determine the 3 year relapse rate defined as time from study entry to induction failure or relapse where deaths or secondary malignancies are competing events.
Treatment-related mortality rate (TRM) | Up to 3 years
  Cumulative incidence estimates will be used to determine the 3 year TRM defined as time from study entry to death where induction failure, relapse or secondary malignancies are competing events.
Number of patients who undergo hematopoietic stem cell transplant (HSCT) | Up to 3 years

OTHER OUTCOMES:
Course duration | Up to 2 years
  Median and range of the length of course duration will be determined.
Length of hospitalization | Up to 2 years
  Median and range of the length of hospitalization time during protocol therapy will be determined.
Time to count recovery | Up to 2 years
  Cumulative incidence estimates that account for competing events will be used to estimate time to count recovery in days where deaths are competing events.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Cooper, Principal Investigator — Children's Oncology Group
Locations (205):
- United States (185):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Leger KJ, Absalon MJ, Demissei BG, Smith AM, Gerbing RB, Alonzo TA, Narayan HK, Hirsch BA, Pollard JA, Razzouk BI, Getz KD, Aplenc R, Kolb EA, Ky B, Cooper TM. Cardiotoxicity of CPX-351 in children and adolescents with relapsed AML: a Children's Oncology Group report. Front Cardiovasc Med. 2024 Jun 14;11:1347547. doi: 10.3389/fcvm.2024.1347547. eCollection 2024. PMID 38947228
- [Derived] Leger KJ, Robison N, Narayan HK, Smith AM, Tsega T, Chung J, Daniels A, Chen Z, Englefield V, Demissei BG, Lefebvre B, Morrow G, Dizon I, Gerbing RB, Pabari R, Getz KD, Aplenc R, Pollard JA, Chow EJ, Tang WHW, Border WL, Sachdeva R, Alonzo TA, Kolb EA, Cooper TM, Ky B. Rationale and design of the Children's Oncology Group study AAML1831 integrated cardiac substudies in pediatric acute myeloid leukemia therapy. Front Cardiovasc Med. 2023 Dec 1;10:1286241. doi: 10.3389/fcvm.2023.1286241. eCollection 2023. PMID 38107263
- [Derived] Andolina JR, Fries C, Boulware R, Vargas A, Fraint E, Barth M, Ambrusko S, Comito M, Monteleone P. Successful Bone Marrow Transplantation With Intensive Post-transplant Intrathecal Chemotherapy for CNS Relapsed AML in 2 Infants. J Pediatr Hematol Oncol. 2022 Jan 1;44(1):e264-e267. doi: 10.1097/MPH.0000000000002151. PMID 33843815